CLINICAL TRIAL: NCT04108065
Title: The Role of Pregnancy-induced Gallbladder Dysmotility in the Pathophysiology of Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-19036095
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; gallbladder motility; glp-1; pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with gestational diabetes mellitus (GDM): GDM diagnosed according to current Danish guidelines (plasma glucose (PG) concentration at 120 min after a 75 g oral glucose tolerance test (OGTT) ≥9.0 mM)
- Pregnant women with normal glucose tolerance (control group): Pregnant women with normal glucose tolerance (fasting plasma glucose (PG) concentration ≤6.0 mM and PG concentration at 120 min after a 75 g-OGTT <7.8 mM)

SUMMARY:
The primary aim of the study is to evaluate postprandial gallbladder emptying and plasma concentrations of the glucose-lowering and satiety-promoting gut hormone glucagon-like peptide 1 (GLP-1) during third trimester of pregnancy in women with gestational diabetes mellitus (GDM) compared with age and body mass index (BMI)-matched pregnant control women with normal glucose tolerance (NGT).

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) defined as glucose intolerance first detected during pregnancy is a strong predictor of future type 2 diabetes. Patients with GDM exhibit severely reduced postprandial responses of the insulinotropic and satiety-promoting gut hormone glucagon-like peptide 1 (GLP-1), which normalise alongside remission of GDM after delivery. Ingested nutrients and bile acids constitute potent stimulators of GLP-1 secretion. Reduced postprandial GLP-1 responses likely contribute to the pathophysiology of GDM, but the mechanisms are unknown. Based on previous studies studying gallbladder emptying during pregnancy, we hypothesize that reduced postprandial GLP-1 responses in GDM is due to incomplete gallbladder emptying during third trimester. If our hypothesis proves right, reduced gallbladder emptying and ensuing attenuation of postprandial GLP-1 secretion will constitute an obvious and druggable target for the treatment of GDM.

Fifteen women with gestational diabetes mellitus and 15 age and body mass index (BMI)-matched pregnant women with normal glucose tolerance will be enrolled in the study. For each subject, the study encompasses one screening visit and two experimental days; one during third trimester of pregnancy and one 3-9 months post partum. On experimental days, a standardised liquid mixed meal test (added 1.5 g of paracetamol for evaluation of gastric emptying according to paracetamol absorption) with repeated ultrasonographic gallbladder scans and blood samples will be performed.

ELIGIBILITY:
Inclusion criteria - women with gestational diabetes mellitus (GDM):

* GDM diagnosed according to current Danish guidelines (plasma glucose (PG) concentration at 120 min after a 75 g oral glucose tolerance test (OGTT) ≥9.0 mM)
* Caucasian ethnicity
* Age >18 years
* Pre-pregnancy BMI <30 kg/m2 and third trimester BMI <35 kg/m2
* Informed oral and written consent

Exclusion criteria - women with gestational diabetes:

* Anaemia (haemoglobin <7.5 mM)
* Previous preeclampsia, HELLP syndrome (haemolysis, elevated liver enzymes and low platelets) and/or pregnancy-induced intrahepatic cholestasis
* Gastrointestinal disease, previous gastric or intestinal resection, cholecystectomy and/or any major intra-abdominal surgery
* Previous pancreatic disease and/or neoplasia
* Postpartum use of hormonal contraception including intrauterine device
* Any condition the investigator group suspect would interfere with trial participation

Inclusion criteria - control group:

* Normal glucose tolerance (fasting plasma glucose (PG) concentration ≤6.0 mM and PG concentration at 120 min after a 75 g-OGTT <7.8 mM)
* Caucasian ethnicity
* Age >18 years
* Pre-pregnancy BMI <30 kg/m2 and third trimester BMI <35 kg/m2
* Informed oral and written consent

Exclusion criteria - control group:

* Anaemia (haemoglobin <7.5 mM)
* Previous preeclampsia, HELLP syndrome (haemolysis, elevated liver enzymes and low platelets) and/or pregnancy induced intrahepatic cholestasis
* Gastrointestinal disease, previous gastric or intestinal resection, cholecystectomy and/or any major intra-abdominal surgery
* Previous pancreatic disease and/or neoplasia
* Postpartum use of hormonal contraception including intrauterine device
* Verified prior GDM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifteen women with gestational diabetes mellitus and 15 age and body mass index (BMI)-matched pregnant women with normal glucose tolerance will be enrolled in the study. Only pregnant women who have been tested for gestational diabetes mellitus will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
GLP-1 response | 240 minutes
  Postprandial GLP-1 response (as assessed by area under curve (AUC) within 240 minutes after meal ingestion) during third trimester compared to 3-9 months postpartum.
Gallbladder emptying | 240 minutes
  Postprandial gallbladder emptying (evaluated as repeated measures of gallbladder volumes using bed-side ultrasonography within 240 minutes after meal ingestion) during third trimester compared to 3-9 months postpartum.

SECONDARY OUTCOMES:
Responses of glucose, insulin, C-peptide, glucagon, GIP | 240 minutes
  Postprandial responses of glucose, insulin, C-peptide, glucagon (as assessed by area under curve (AUC) during third trimester compared to 3-9 months postpartum.
Gastric emptying | 240 minutes
  Postprandial responses of paracetamol (as assessed by area under curve (AUC) during third trimester compared to 3-9 months postpartum.
Bile acid and gallbladder physiology | 240 minutes
  Postprandial responses of GLP-2, CCK, total bile acids, C4 and FGF-19 (as assessed by area under curve (AUC) during third trimester compared to 3-9 months postpartum.
Oxytocin | 240 minutes
  Postprandial responses of oxytocin (as assessed by area under curve (AUC) during third trimester compared to 3-9 months postpartum.
GDF15 | 240 minutes
  Postprandial responses of GDF-15 (as assessed by area under curve (AUC) during third trimester compared to 3-9 months postpartum.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No